CLINICAL TRIAL: NCT03820323
Title: Optimizing Viral Load Suppression in Kenyan Children on Antiretroviral Therapy
Acronym: Opt4Kids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Kenya Medical Research Institute (Other); University of Colorado, Denver (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Rena Patel, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: STUDY000004861; R34MH115769 (NIH)
Record Dates: First submitted 2019-01-23; First posted 2019-01-29 (Actual); Results first posted 2022-12-27 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Chronic HIV Infection

STUDY DESIGN:
Intervention Model Description: Randomized control trial of two study arms
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and those conducting the analysis will be blinded to arm allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Other): Participants in the Standard-of-Care control arm will receive laboratory based VL testing based on the existing Kenyan national guidelines by routine clinical staff (not study staff). DRM testing is usually done if there is a failing 2nd line ART regimen based on the current Kenyan guideline.
  Interventions: Diagnostic Test: SOC VL testing
- Intervention (Experimental): POC VL and targeted DRM testing.
  Interventions: Diagnostic Test: POC VL and targeted DRM testing.

INTERVENTIONS:
Diagnostic Test: POC VL and targeted DRM testing. — Point-of-care Viral Load Testing will be done to ensure that providers and caregivers receive the results with in 24 hours study. Targeted DRM testing will be performed during the initiation of ART and when viremia (VL>1000 copies/mL) is detected.
  Arms: Intervention
Diagnostic Test: SOC VL testing — SOC VL testing is done at 6 months after ART initiation then every 3 months if unsuppressed, otherwise every 12 months. DRM testing is conducted only if failing 2nd line ART.
  Other Names: Kenyan National guidelines for viral load testing
  Arms: Standard of Care

SUMMARY:
Among nearly 1 million HIV-infected children receiving antiretroviral treatment (ART), as many as 40% of those living in resource limited settings have not achieved virologic suppression. Kenya, a The Joint United Nations Programme on HIV/AIDS (UNAIDS) fast-track and The U.S. President's Emergency Plan for AIDS Relief (PEPFAR) priority country, has an estimated 98,000 children aged 0-14 years living with HIV. Virologic suppression is achieved by only 65% of Kenyan children on ART translating to only 38% of the final UNAIDS 90-90-90 goal for population-level viral suppression. Feasible, scalable and cost-effective approaches to maximizing durability of first-line ART and ensuring viral load (VL) suppression in HIV-infected children are urgently needed. This pilot study will evaluate two critical components related to viral suppression in children via: 1) Point-of-care (POC) VL testing (Aim 1) and 2) targeted drug resistance mutation (DRM) testing (Aim 2) among children on first-line ART at three facilities within a PEPFAR-funded HIV care and treatment program in Kenya. The hypotheses are: 1) viral suppression rates will be higher among children with access to POC VL testing and time to suppression shorter compared to children with standard VL testing and 2) DRM testing will shorten time to viral suppression and that the investigators will observe high levels of 1st line antiretroviral DRMs among children on ART without viral suppression. This proposal directly addresses the urgent need to find interventions to maximize viral suppression among children on ART and achieve the UNAIDS 90-90-90 goals.

DETAILED DESCRIPTION:
The study design will be a randomized, controlled study to pilot the use of POC VL and DRM testing in children aged 1-14 years on first-line ART. Children enrolling at each site will be randomized 1:1 to two study arms.

Standard of Care Arm:

Participants in the Standard-of-Care (SOC) control arm will receive the standard-of-care VL and DRM testing based on the existing Kenyan national guidelines. VL testing will be 6 months after ART initiation (then every 3 months if unsuppressed, otherwise every 12 months) with DRM testing only if failing second-line ART. Children who have a high lab-based HIV VL (≥1,000 copies/mL) will receive intensive adherence counseling and be asked to return to the clinic in 3 months for repeat HIV VL testing. If the HIV VL remains high (≥1,000 copies/mL), the children will be managed per Kenya national guidelines.

Intervention Arm:

Children in the intervention arm will undergo POC VL testing every 3 months for a total of 12 months. "Targeted" DRM testing will include DRM testing for each child on the first detection of lack of viral suppression (VL > 1000 copies/mL) and in children newly initiating ART.

The investigators will follow the viral outcomes 12 months after the implementation of POC VL testing and compare VL suppression rates, defined as VL <1000 copies/mL by the Kenyan national guidelines, among intervention vs. control arms, accounting for pre-intervention VL suppression rates.

The primary outcome for Aim 1 is rates of viral suppression (defined as VL <1000 copies/mL) at 12 months after POC VL testing implementation at the three facilities. The secondary outcome for Aim 1 is time to viral suppression among those children without viral suppression at their 1st POC VL testing or newly initiating ART after POC VL testing implementation. In Aim 2, the investigators intend to evaluate the impact of targeted HIV DRM testing on viral suppression in the intervention arm only. The investigators will also explore how sociodemographic, behavioral, clinical, and facility factors may be contributing to the DRM patterns they observe.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-14 years living with HIV (documented HIV positive)
* On first-line ART per Kenyan National Guideline or
* Newly initiating ART

Exclusion Criteria:

* On second-line, third-line, or non-standard first-line ART

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 704 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rena Patel, MD, MPH, Principal Investigator — University of Alabama at Birmingham; Lisa L Abuogi, MD, MSc, Principal Investigator — University of Colorado, Denver
Locations (1):
- Rtcp-Faces, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all outcome measures will be made available after study completion
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After primary outcomes results are published.
Access Criteria: Contact PIs of the study and obtain institutional ethic review approvals.

REFERENCES:
- [Derived] Scallon AJ, Hassan SA, Qian SR, Gao Y, Oyaro P, Brown E, Wagude J, Mukui I, Kinywa E, Oluoch F, Odhiambo F, Oyaro B, Kingwara L, Yongo N, Karauki E, Otieno L, John-Stewart GC, Abuogi LL, Patel RC. "I feel drug resistance testing allowed us to make an informed decision": qualitative insights on the role of HIV drug resistance mutation testing among children and pregnant women living with HIV in western Kenya. BMC Health Serv Res. 2023 Aug 24;23(1):908. doi: 10.1186/s12913-023-09804-x. PMID 37620855
- [Derived] Qian SRW, Hassan SA, Scallon AJ, Oyaro P, Brown E, Wagude J, Mukui I, Kinywa E, Oluoch F, Odhiambo F, Oyaro B, Kingwara L, Yongo N, Karauki E, Gao J, Otieno L, John-Stewart GC, Abuogi LL, Patel RC. "After viral load testing, I get my results so I get to know which path my life is taking me": qualitative insights on routine centralized and point-of-care viral load testing in western Kenya from the Opt4Kids and Opt4Mamas studies. BMC Health Serv Res. 2022 Dec 17;22(1):1540. doi: 10.1186/s12913-022-08593-z. PMID 36528677
- [Derived] Patel RC, Oyaro P, Thomas KK, Wagude J, Mukui I, Brown E, Hassan SA, Kinywa E, Oluoch F, Odhiambo F, Oyaro B, Kingwara L, Karauki E, Yongo N, Otieno L, John-Stewart GC, Abuogi LL. Point-of-care HIV viral load and targeted drug resistance mutation testing versus standard care for Kenyan children on antiretroviral therapy (Opt4Kids): an open-label, randomised controlled trial. Lancet Child Adolesc Health. 2022 Oct;6(10):681-691. doi: 10.1016/S2352-4642(22)00191-2. Epub 2022 Aug 18. PMID 35987208
- [Derived] Patel RC, Oyaro P, Odeny B, Mukui I, Thomas KK, Sharma M, Wagude J, Kinywa E, Oluoch F, Odhiambo F, Oyaro B, John-Stewart GC, Abuogi LL. Optimizing viral load suppression in Kenyan children on antiretroviral therapy (Opt4Kids). Contemp Clin Trials Commun. 2020 Oct 27;20:100673. doi: 10.1016/j.conctc.2020.100673. eCollection 2020 Dec. PMID 33195874

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Kisumu County, western Kenya, with the second-highest prevalence of pediatric HIV infections in Kenya. The study was implemented at five low-resource, high-HIV burden public sector facilities from March 2019 to December 2020. We chose the study facilities to leverage existing POC technologies, specifically the GeneXpert® platform.
Period: Overall Study
Arm/Group | Standard of Care | Intervention
Started | 355 | 349
Completed | 315 | 313
Not Completed | 40 | 36
Not completed — Lost to Follow-up | 2 | 1
Not completed — Missed 12-month visit | 22 | 14
Not completed — Death | 2 | 1
Not completed — Transferred out | 13 | 11
Not completed — Terminated | 0 | 3
Not completed — Withdrawal by Subject | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Intervention | Total
Number analyzed (Participants) | 355 | 349 | 704
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 355 | 349 | 704
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 9 [7 to 12] | 9 [6 to 12] | 9 [7 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 184 | 344
  Male | 195 | 165 | 360
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 355 | 349 | 704
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 355 | 349 | 704
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 355 | 349 | 704
Virological suppression at enrollment [Count of Participants; unit: Participants] — Viral load <1000 copier per mL at enrollment or most recent up to 2 years prior
  Participants
    Yes (viral load <1000 copies per mL) | 274 | 262 | 536
    No (viral load >=1000 copies per mL) | 39 | 38 | 77
    No viral load recorded or missing | 42 | 49 | 91

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Viral Suppression
Description: Viral Load <1000 copies/mL at 12 months after enrollment
Time Frame: 12 months after enrollment
Measure: Number; unit: participants
Groups:
- Standard of Care: Participants in the Standard-of-Care (SOC) control arm will receive laboratory based viral load (VL) testing based on the existing Kenyan national guidelines by routine clinical staff (not study staff). Drug resistance mutation (DRM) testing is usually done if there is a failing 2nd line antiretroviral therapy (ART) regimen based on the current Kenyan guideline.
  SOC VL testing: SOC VL testing is done at 6 months after ART initiation then every 3 months if unsuppressed, otherwise every 12 months. DRM testing is conducted only if failing 2nd line ART.
- Intervention: Point-of-care (POC) viral load (VL) and targeted Drug resistance mutation (DRM) testing.
  POC VL and targeted DRM testing: POC VL testing will be done to ensure that providers and caregivers receive the results with in 24 hours study. Targeted DRM testing will be performed during the initiation of antiretroviral (ART) and when viremia (VL>1000 copies/mL) is detected.
Arm/Group | Standard of Care | Intervention
Number analyzed (Participants) | 315 | 313
participants | 289 | 283
Statistical Analysis 1: Comparison: Standard of Care vs Intervention; Test type: Superiority; p = 0.55, Modified Poisson regression; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.94 to 1.03]

2. Secondary Outcome: Virological Suppression at 12 Months Among Children Newly Initiating ART or Initially Virologically Unsuppressed
Description: Among children newly initiating ART or initially virologically unsuppressed, we then evaluated the virological suppression status at 12 months post-enrollment.
Time Frame: 12 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Intervention
Number analyzed (Participants) | 59 | 60
Participants | 42 | 36
Statistical Analysis 1: Comparison: Standard of Care vs Intervention; Test type: Superiority; p = 0.28, Modified Poission regression; Risk Ratio (RR) = 0.86, 95% CI 2-sided [0.66 to 1.13]

3. Secondary Outcome: Number of Participants Who Underwent POC VL Testing
Description: The number of children undergoing VL testing within each group (POC VL testing or SOC VL testing) at the scheduled intervals.
Time Frame: Every 3 months within the 12 months study period
Population: Of note, during the 6- and 9-month study visits, COVID-19 related restrictions in travel and routine care greatly affected our ability to obtain samples for VL testing leading to varying numbers analyzed per month.
Measure: Number; unit: participants
Arm/Group | Standard of Care | Intervention
Number analyzed (Participants) | 355 | 349
participants
  0 months: number analyzed (Participants) | 351 | 349
  0 months | 167 | 349
  3 months: number analyzed (Participants) | 351 | 329
  3 months | 185 | 301
  6 months: number analyzed (Participants) | 351 | 321
  6 months | 131 | 177
  9 months: number analyzed (Participants) | 351 | 335
  9 months | 143 | 186
  12 months: number analyzed (Participants) | 351 | 286
  12 months | 135 | 286

4. Secondary Outcome: Turn-around Time for the VL Testing Results
Description: The time it takes for viral load results to be received by health care providers and participants.
Time Frame: Every 3 months within the 12 months study period
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Standard of Care | Intervention
Number analyzed (Participants) | 355 | 349
days | 15 [10 to 21] | 1 [0 to 1]

5. Secondary Outcome: Number of Children With Any or Major Drug Resistance Mutations (DRMs)
Description: The number of children tested for DRMs with any or major mutations within each class of HIV drugs.
Time Frame: 12 months post enrollment
Population: Of 120 samples in the intervention group in which we requested a DRM test, 13 (11%) failed to amplify. We are not able to elucidate reasons why five of the samples in the Standard of Care group were selected for DRM testing or why three of the five requested DRM tests were not performed successfully.
Measure: Number; unit: participants
Arm/Group | Standard of Care | Intervention
Number analyzed (Participants) | 2 | 107
participants
  Any DRM | 2 | 107
  NRTI | 1 | 61
  NNRTI | 2 | 88
  Protease Inhibitor | 1 | 9
  Any major DRM | 2 | 91
  Major NRTI | 1 | 61
  Major NNRTI | 2 | 88
  Major protease Inhibitor | 1 | 9

ADVERSE EVENTS:
Time Frame: The adverse events were reported from enrollment to approximately 12 months after enrollment for each participant.
Arm/Group | Standard of Care | Intervention
All-Cause Mortality (participants affected / at risk) | 2/355 | 1/349
Serious Adverse Events (participants affected / at risk) | 1/355 | 0/349
Other Adverse Events (participants affected / at risk) | 0/355 | 0/349
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (N=355) | Intervention (N=349)
Hospitalization (Gastrointestinal disorders) | 1 (1) | NA — Malnutrition

LIMITATIONS AND CAVEATS:
First, it is possible we had sample biased towards higher levels of viral suppression (VS). Second, though our package of POC VL testing, DRM testing, and clinical decision support was only offered to intervention group, the same providers cared for participants in intervention and control groups. Third, VS was assessed on different schedules for intervention and control, the intervention group participants had a greater number of opportunities to act on their test results and detect viremia.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT03820323/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT03820323/SAP_001.pdf